CLINICAL TRIAL: NCT04606381
Title: An Open-label, Multicenter, Dose Escalation Phase 1b Study to Assess the Safety and Pharmacokinetics of Subcutaneous Delivery of Amivantamab, a Human Bispecific EGFR and cMet Antibody for the Treatment of Advanced Solid Malignancies
Brief Title: A Study of Amivantamab Subcutaneous (SC) Administration for the Treatment of Advanced Solid Malignancies
Acronym: PALOMA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108891; 61186372NSC1003 (Other: Janssen Research & Development, LLC); 2020-003225-36 (EudraCT Number)
Record Dates: First submitted 2020-10-06; First posted 2020-10-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
Keywords: Amivantamab; JNJ-61186372
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Ami-LC-MD and Ami-LC (Experimental): Participants in cohort 1a will receive amivantamab admixed with rHuPH20 (Ami-LC-MD) subcutaneous (SC) infusion and participants in cohort 1b will receive amivantamab (Ami-LC) SC infusion.
  Interventions: Drug: Ami-LC-MD; Drug: Ami-LC
- Part 2: Ami-HC and Ami-HC-CF (Experimental): Participants will receive SC infusion of newly developed high concentration amivantamab (Ami-HC) or SC injection of amivantamab co-formulated with rHuPH20 (Ami-HC-CF).
  Interventions: Drug: Ami-HC; Drug: Ami-HC-CF

INTERVENTIONS:
Drug: Ami-LC-MD — Participants will receive amivantamab admixed with rHuPH20 SC infusion.
  Arms: Part 1: Ami-LC-MD and Ami-LC
Drug: Ami-LC — Participants will receive amivantamab SC infusion.
  Arms: Part 1: Ami-LC-MD and Ami-LC
Drug: Ami-HC — Participants will receive amivantamab SC infusion.
  Arms: Part 2: Ami-HC and Ami-HC-CF
Drug: Ami-HC-CF — Participants will receive amivantamab co-formulated with rHuPH20 as SC injection.
  Arms: Part 2: Ami-HC and Ami-HC-CF

SUMMARY:
The purpose of this study is to assess the feasibility of subcutaneous (SC) administration of amivantamab based on safety and pharmacokinetics and determine a dose, dose regimen and formulation for amivantamab SC delivery.

ELIGIBILITY:
Inclusion criteria:

* Part 1 and Part 2: Participant must have histologically or cytologically confirmed solid malignancy that is metastatic or unresectable and which may derive benefit from epidermal growth factor receptor (EGFR) or mesenchymal-epidermal transition tyrosine kinase receptor/hepatocyte growth factor receptor (cMet) directed therapy. Eligible tumor types include non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), hepatocellular cancer (HCC), colorectal cancer (CRC), renal cell cancer (RCC), medullary thyroid cancer (MTC), gastroesophageal cancer (GEC), mesothelioma, breast cancer (BC) and ovarian cancer (OC). Participants must have either progressed after prior standard of care therapy for metastatic disease, be ineligible for, or have refused all other currently available therapeutic options. In cases where participants refuse currently available therapeutic options, this must be documented in the study records.
* Participant must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at Screening and a negative urine or serum pregnancy test within 24 hours before the first dose of study drug
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study drug
* A man who is sexually active with a woman of childbearing potential must agree to use a condom and his partner must also be practicing a highly effective method of contraception (that is, established use of oral, injected or implanted hormonal methods of contraception; placement of an Intrauterine device [IUD] or Intrauterine system [IUS])

Exclusion criteria:

* Participant has uncontrolled inter-current illness, including but not limited to poorly controlled hypertension or diabetes, ongoing or active systemic infection (that is, has discontinued all antibiotics for at least one week prior to first dose of study drug), diagnosed or suspected viral infection (except Human immunodeficiency virus [HIV] positive participants with 1 or more of the following: a) not receiving highly active antiretroviral therapy; b) a change in antiretroviral therapy within 6 months of the start of screening; c) cluster of differentiation 4 (CD4)+ T-cell count less than [<]350 per cubic millimeters [mm^3] at screening; d) an acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening), or psychiatric illness/social situation that would limit compliance with study requirements, including ability to self-care for anticipated toxicities [that is. rash or paronychia]. Participants with medical conditions requiring chronic continuous oxygen therapy are excluded
* Participant has had prior chemotherapy, targeted cancer therapy, or treatment with an investigational anti-cancer agent within 2 weeks or 4 half-lives, whichever is longer, before the first administration of study drug; or participant has received prior immunotherapy within 6 weeks before the first administration of study drug. For agents with long half-lives, the maximum required time since last dose is 4 weeks. Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less, (except for alopecia [any grade], Grade less than or equal to [<=] 2 peripheral neuropathy, and Grade less than [<] 2 hypothyroidism stable on hormone replacement). Autoimmune toxicities from previous immunotherapy must be fully resolved to baseline levels
* Participants with untreated brain metastases. Participants with locally treated metastases that are clinically stable and asymptomatic for at least 2 weeks and who are off or receiving low-dose corticosteroid treatment (<=10 milligrams [mg] prednisone or equivalent) for at least 2 weeks prior to study treatment are eligible
* Participant has an active malignancy other than the disease under study requiring treatment
* Participant has leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Observed Amivantamab Serum Concentration Immediately Prior to the Next Dose Administration (Ctrough) | Up to Day 29
  Ctrough is the observed amivantamab serum concentration immediately prior to the next drug administration.
Number of Participants with Adverse Event (AE) | Up to 4 years 1 month
  An adverse event is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An adverse event does not necessarily have a causal relationship with the drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Number of Participants with Dose Limiting Toxicity (DLT) | Up to Day 28
  Number of participants with DLT will be assessed.
Number of Participants with Clinical Laboratory Abnormalities | Up to 4 years 1 month
  Number of participants with clinical laboratory (hematology, clinical chemistry, and urinalysis) abnormalities will be assessed.

SECONDARY OUTCOMES:
Number of Participants with Anti-amivantamab and Anti-rHuPH20 antibodies | Up to 4 years 1 month
  Number of participants with anti-amivantamab and anti-rHuPH20 antibodies will be assessed.
Epidermal Growth Factor Receptor (EGFR) Concentrations | Up to 4 years 1 month
  EGRF concentrations markers will be assessed.
Mesenchymal-Epidermal Transition Tyrosine Kinase Receptor/Hepatocyte Growth Factor Receptor (cMET) Markers | Up to 4 years 1 month
  cMET markers will be analyzed.
Overall Response Rate (ORR) | Up to 4 years 1 month
  ORR defined as the proportion of participants with partial response (PR) or better according to Response Criteria in Solid Tumors (RECIST) v1.1.
Part 2: Maximum Amivantamab Dosing Interval Between Time Zero to Steady State | Up to 4 years 1 month
  Maximum amivantamab dosing interval Between time zero to steady state will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (12):
- United States (5):
  - Cedars Sinai Medical Center, West Hollywood, California
  - Community Health Network, Indianapolis, Indiana
  - Langone Health at NYC University, NYU School of Medicine, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
- University Health Network, Toronto, Ontario, Canada
- South Korea (4):
  - Chungbuk National University Hospital, Cheongju-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- United Kingdom (2):
  - The Christie Nhs Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency